CLINICAL TRIAL: NCT05055570
Title: The Mechanism Research of Angiotensin II Pathway and Postoperative Hypoxemia
Brief Title: Angiotensin II Pathway and Postoperative Hypoxemia
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Jun Ma, The chief of department of anesthesiology, Beijing Anzhen Hospital
Other Study IDs: 2021107X
Record Dates: First submitted 2021-09-07; First posted 2021-09-24 (Actual); Results first posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-04

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoxemia group: oxygenation index (OI)≤200
  Interventions: Other: No intervention
- Non-hypoxemia group: oxygenation index (OI)>200
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Acute type A aortic dissection is often accompanied by postoperative hypoxemia, the cause of which is not fully understood. Angiotensin II is an important component of the renin-angiotensin system (RAS), which has been suggested to be involved in the development of aortic dissection and pulmonary inflammation.The purpose of this study was to investigate the role and mechanism of angiotensin II pathway in postoperative hypoxemia after acute type A aortic dissection, and to provide reference for clinical application

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery for acute type A aortic dissection
* age between 18 to 80

Exclusion Criteria:

* perioperative severe cardiac insufficiency
* rejection of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical treatment for acute type A aortic dissection in our hospital were selected. The age was 18 years ≤ age ≤80years, and gender was not limited. The overall study patients were divided into the hypoxemia group and non-hypoxemia group according to the presence or lack of hypoxemia after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Anzhen hospital, Beijing, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang X, Ma J, Lin D, Dong X, Wu J, Bai Y, Zhang D, Gao J. The risk factors of postoperative hypoxemia in patients with Stanford type A acute aortic dissection. Medicine (Baltimore). 2023 Aug 18;102(33):e34704. doi: 10.1097/MD.0000000000034704. PMID 37603505

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypoxemia Group | Non-hypoxemia Group
Started | 25 | 63
Completed | 25 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypoxemia Group | Non-hypoxemia Group | Total
Number analyzed (Participants) | 25 | 63 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.6) | 50.4 (10.5) | 50.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 19 | 27
  Male | 17 | 44 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 63 | 88
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kg] | 83.9 (14.9) | 74.4 (12.8) | 77.1 (14.0)
Hight [Mean (Standard Deviation); unit: cm] | 169.7 (7.6) | 171.6 (8.9) | 171.1 (8.6)
BMI [Mean (Standard Deviation); unit: kg / m2] | 29.0 (3.7) | 25.2 (3.4) | 26.3 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: The Difference Concentrations of ANG II in Serum Between Patients With and Without Postoperative Hypoxemia.
Description: Blood samples were taken within 24 hours after operation to detect the contents of ANG II in serum. Postoperative hypoxemia is defined by the oxygenation index (OI), which is the ratio of arterial partial pressure of oxygen to fraction inspired oxygen (PaO2 / FiO2), of less than or equal to 200 for two consecutive times within the first 24 h after operation
Time Frame: Within 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: pg / mL
Groups:
- Hypoxemia Group: oxygenation index （PaO2 / FiO2）≤200
- Non-hypoxemia Group: oxygenation index （PaO2 / FiO2）>200
Arm/Group | Hypoxemia Group | Non-hypoxemia Group
Number analyzed (Participants) | 25 | 63
pg / mL | 100 [73.9 to 117.6] | 78.5 [60.9 to 92.1]

2. Secondary Outcome: The Risk Factors for Postoperative Hypoxemia in Stanford Type A Acute Aortic Dissection Patients.
Description: Basic characteristics, intraoperative details, biochemical parameters and outcome results were obtained, and blood was collected within 24 hours after surgery for the measurement of ANG II, sACE2 and mir-145 concentrations. Univariate analysis was first performed to identify the potential risk factors for postoperative hypoxemia. Multivariate logistic regression analysis was performed for factors with P < 0.05 or that were considered clinically important.
Time Frame: up to 60 days
Reporting Status: Not Posted

3. Secondary Outcome: Duration of Stay in the Intensive Care Unit
Description: Duration of Stay in the intensive care unit after surgery
Time Frame: up to 60 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One month after surgery
Arm/Group | Hypoxemia Group | Non-hypoxemia Group
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/63
Other Adverse Events (participants affected / at risk) | 0/25 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT05055570/Prot_SAP_000.pdf